CLINICAL TRIAL: NCT00048789
Title: Treatment of Chronic Graft Versus Host Disease With Extracorporeal Photopheresis
Brief Title: Extracorporeal Photopheresis to Treat Chronic Graft-Versus-Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030025; 03-I-0025
Record Dates: First submitted 2002-11-07; First posted 2002-11-08 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-01-29

CONDITIONS: Graft vs Host Disease
Keywords: Psoralen; Refractory; Transplantation; Stem Cell; UVA; Graft-versus-host Disease; GVHD
MeSH Terms: conditions — Graft vs Host Disease | interventions — Photopheresis

INTERVENTIONS:
Procedure: Extracorporeal Photopheresis

SUMMARY:
This study will examine the safety and effectiveness of extracorporeal photopheresis (ECP) for treating chronic graft-versus-host disease (GvHD). GvHD is a common complication of stem cell transplantation using donated stem cells. It occurs when the donor's T-lymphocytes (a type of immune cell) see the patient's cells as foreign and mount an immune response to reject them. The attack can cause skin rash, mouth sores, liver or lung inflammation, lack of appetite, and muscle stiffness. Chronic GvHD can cause serious illness, and even death, from the long-term effects of immune dysfunction and from toxic effects of medications (such as cyclosporine and prednisone) used to treat it.

ECP is an experimental treatment designed to stop the lymphocytes from attacking the body. It involves collecting some of the cells that cause GvHD, treating them with a combination of drug and light therapy and returning them to the body. Sixty to 80 percent of patients with chronic GvHD improve with ECP treatment, and some patients can stop treatment with prednisone or cyclosporine, or reduce the drug dosages.

Patients with chronic GvHD whose condition has not improved after a minimum 14-day course of cyclosporine and prednisone may be eligible for this study. Patients must be able to travel to the NIH Clinical Center in Bethesda, Maryland, twice a week during the 3-month study period.

Upon entering the study, participants will have a baseline evaluation to measure the extent of GvHD. This assessment includes blood tests, eye and dental examinations, skin biopsy for patients with skin involvement, and CT scans and lung function tests to look for possible lung involvement. Biopsies of the lung, liver, mouth, or eye may be requested if needed to confirm GvHD in these tissues. The skin will be photographed before starting ECP treatment and once a month during the treatment period. Following baseline tests, participants will undergo treatment and evaluations as follows:

ECP Treatment

Patients will have blood drawn to collect lymphocytes causing GvHD. This may be done with a special needle or catheter (tube inserted into a vein) or for patients who need or prefer it with a temporary central venous catheter similar to that used for the stem cell transplantation. Patients will have three 2- to 3-hour treatments a week for the first week and two treatments a week after that for a total of 25 treatments over 3 months. Patients who do not tolerate the treatment...

DETAILED DESCRIPTION:
This is a phase 2 study of extracorporeal photopheresis (ECP) for treatment of chronic graft versus host disease following allogeneic hematopoietic stem cell transplantation. Extracorporeal exposure of human mononuclear cells to ultraviolet A radiation following photosensitization with 8-methoxypsoralen has proven to be an effective treatment for cutaneous T-cell lymphoma. Small, single institution studies have suggested efficacy in other T-cell mediated diseases such as solid organ rejection and graft versus host disease. This a phase 2 study of ECP for treatment of chronic graft versus host disease. Eligible patients must have objective evidence of chronic graft versus host disease that is refractory to conventional therapy or must have steroid-dependent disease that does not permit steroid dose reduction. The primary objective of this study is to better define the safety, efficacy and mechanism of action of ECP for treatment of patients with chronic graft versus host disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Objective evidence of chronic graft versus host disease involving the skin, lungs, gastrointestinal tract, liver, or eyes.
  2. Progressive or stable GvHD despite a minimum of 30 days treatment with a calcineurin inhibitor (cyclosporine or tacrolimus) at therapeutic plasma levels, plus at least one other another agent with a different mechanism of action used concurrently for at least 30 days at doses known to be therapeutic for cGvHD. In most cases this second agent will be a corticosteroid administered either as high level pulse dosing (greater than or equal to mg/kg/day prednisone or equivalent in pulses of 3 days or longer for at least two occasions during the qualifying 30 days) and/or daily dosing (greater than or equal to 0.25mg/kg) or alternate day dosing (greater than or equal to 0.50 mg/kg) prednisone or equivalent. In other cases where use of steroids is medically undesirable or contraindicated, the second agent may be mycophenolate mofetil, sirolimus, hydroxychloroquine, clofazimine, thalidomide, azathioprine, pentostatin, etanercept, Infliximab, Rituximab or Daclizumab used at doses and schedule known to provide benefit to patients with cGvHD. Patients in whom calcineurin inhibitors are medically contraindicated may also be eligible for enrollment if there has been at least a 30 day trial of prednisone (or equivalent) at the doses/schedules noted above plus one of the second agents listed above. Patients in whom both calcineurin inhibitors and steroids are medically contraindicated or in whom these agents can be used at only limiting doses may also be eligible if at least two of the alternate agents noted above have been tried for 30 days without further improvement in symptoms of cGvHD. Patients who have stabilization of disease on calcineurin inhibitors plus steroids (or the other combinations noted above), but in whom these medications cannot be tapered without disease flare are also eligible.
  3. Adequate (as determined by PI) renal, hepatic, and cardiac reserve to enable the patient to tolerate Extracorporeal Photopheresis.
  4. The patient's malignancy (if applicable) is in complete remission or the patient is not a candidate for further immune-based anti-tumor therapy (such as donor lymphocyte infusions or immunomodulatory cytokines) due to severity of GvHD.
  5. WBC greater than or equal to 1000 and platelets greater than or equal to 25,000.
  6. Weight greater than or equal to 30kg.
  7. Female patients not pregnant and agree to use a reliable method of birth control during the treatment period
  8. Systolic blood pressure greater than or equal to 90 mm Hg.
  9. Karnofsky score or Lansky score greater than or equal to 30.
  10. Predicted life expectancy of at least 3 months.
  11. A minimum of 100 days following stem cell transplantation.
  12. A minimum of 30 days without a response to, and 7 days following cessation of, certain investigational 2nd-line agents for treatment of GvHD (specifically: thalidomide, azathioprine, pentostatin, etanercept, Infliximab, Rituximab or Daclizumab).
  13. History of failure to achieve any clinical benefit from a previous treatment with ECP where at least 3 months (12 weeks) of twice a week every other week therapy was administered.
  14. Signed and witnessed informed consent.
  15. Hemoglobin greater than 9.5, hematocrit greater than 28.5 (patients not meeting this inclusion criterion may be treated with iron supplementation and/or erythropoietin/darbepoetin until their hgb/hct are in the Inclusion range and may then be reconsidered for study entry).

EXCLUSION CRITERIA:

1. Hypersensitivity or allergy to psoralen (methoxypsoralen).
2. Hypersensitivity to both heparin and/or citrate products.
3. Patients who are unable to visit the NIH clinical center twice a week for at least the first four week treatment period of ECP treatments; or for the NIH or arranged home treatments with ECP thereafter; or for the every 4 week medical evaluation visits to NIH.
4. Frank gastrointestinal bleeding due to GvHD (occult blood positivity excluded).
5. Patients taking a cancer chemotherapeutic agent for continued treatment of malignancy.
6. Patients undergoing radiation therapy.
7. The patient's malignancy (if applicable) is NOT in complete remission or the patient is a candidate for further immune-based anti-tumor therapy (such as donor lymphocyte infusions or immunomodulatory cytokines) to treat GvHD.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 2002-11-04; Study Completion 2009-01-29

PRIMARY OUTCOMES:
Determination of response rate including degree of improvement; steroid sparing effect; types of cGVHD problems which respond to this therapy; assessment of problems or side effects or adverse events associated with the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Akpek G, Zahurak ML, Piantadosi S, Margolis J, Doherty J, Davidson R, Vogelsang GB. Development of a prognostic model for grading chronic graft-versus-host disease. Blood. 2001 Mar 1;97(5):1219-26. doi: 10.1182/blood.v97.5.1219. PMID 11222363
- [Background] Sullivan KM, Witherspoon RP, Storb R, Deeg HJ, Dahlberg S, Sanders JE, Appelbaum FR, Doney KC, Weiden P, Anasetti C, et al. Alternating-day cyclosporine and prednisone for treatment of high-risk chronic graft-v-host disease. Blood. 1988 Aug;72(2):555-61. PMID 3042042
- [Background] Yoo EK, Rook AH, Elenitsas R, Gasparro FP, Vowels BR. Apoptosis induction of ultraviolet light A and photochemotherapy in cutaneous T-cell Lymphoma: relevance to mechanism of therapeutic action. J Invest Dermatol. 1996 Aug;107(2):235-42. doi: 10.1111/1523-1747.ep12329711. PMID 8757769